CLINICAL TRIAL: NCT06301165
Title: TPC Versus GP Induction Chemotherapy Followed by Concurrent Chemoradiotherapy for High-risk Locoregionally Advanced Nasopharyngeal Carcinoma, a Multi-center Phase II Randomized Trial
Brief Title: TPC Versus GP Induction Chemotherapy for Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-FXY-129
Record Dates: First submitted 2024-02-24; First posted 2024-03-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Polymeric micellar paclitaxel; TPC; GP
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPC induction chemotherapy + CCRT (Experimental): TPC induction chemotherapy regimen followed by concurrent chemoraditherapy (cisplatin 100 mg/m2, every 3 weeks for 3 cycles) and IMRT (PTVnx 70Gy/33f; PTVnd 70Gy/33f; PTV1 60Gy/33f; PTV2 54Gy/33f)
  Interventions: Drug: TPC induction chemotherapy
- GP induction chemotherapy + CCRT (Active Comparator): GP induction chemotherapy regimen followed by concurrent chemoraditherapy (cisplatin 100 mg/m2, every 3 weeks for 3 cycles) and IMRT (PTVnx 70Gy/33f; PTVnd 70Gy/33f; PTV1 60Gy/33f; PTV2 54Gy/33f)
  Interventions: Drug: GP induction chemotherapy

INTERVENTIONS:
Drug: TPC induction chemotherapy — TPC induction chemotherapy regimen contains Polymeric micellar paclitaxel, which is a novel Cremophor EL-free, nanoparticle micellar formulation of paclitaxel, cisplatin and capecitabine. TPC induction chemotherapy regimen (polymeric micellar paclitaxel 200 mg/m2 D1, cisplatin 75 mg/m2 D1, capecitabine 1000 mg/m2/day D1-14, every 3 weeks for 3 cycles).
  Arms: TPC induction chemotherapy + CCRT
Drug: GP induction chemotherapy — GP induction chemotherapy regimen (gemcitabine 1000 mg/m2 D1/8, cisplatin 80 mg/m2 D1, every 3 weeks for 3 cycles)
  Arms: GP induction chemotherapy + CCRT

SUMMARY:
The NCCN guidelines recommend induction chemotherapy followed by concurrent chemoradiotherapy as the standard treatment for locoregionally advanced nasopharyngeal carcinoma (NPC). However, meta-analyses have shown significant survival differences between different induction chemotherapy regimens. How to choose an induction chemotherapy regimen and treatment course that ensures definitive therapeutic effects and low incidence of toxic side effects remains a hot spot in clinical research. Polymeric micellar paclitaxel are an innovative form of paclitaxel drugs, with high penetration and long retention effects, which can enter the vascularly disordered tumor microenvironment through passive targeting and form higher concentrations in tumor tissue. It remains to be investigated whether the TPC (paclitaxel, cisplatin and capecitabine) regimen based on polymeric micellar paclitaxel compared to the current standard first-line induction chemotherapy GP (gemcitabine, cisplatin) regimen can further improve therapeutic effects in high-risk patients with locally advanced disease. There is still a lack of head-to-head studies for comparison. This study aims to compare, through a prospective, parallel-controlled, randomized, open-label, multicenter phase II clinical trial, the TPC induction chemotherapy vs. the GP induction chemotherapy combined with concurrent chemoradiotherapy for the treatment of high-risk locoregionally advanced NPC (T4 or N2-3) in terms of 2-year progression-free survival, overall survival, overall response rate, toxic side effects, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years;
2. Pathologically confirmed differentiated non-keratinizing carcinoma and undifferentiated non-keratinizing carcinoma (WHO type II or III);
3. Staged as T4N0-3M0 or T1-4N2-3M0 (UICC 8th edition);
4. Easte Cooperative Oncology Group performance status of 0 or 1;
5. Adequate bone marrow: leucocyte count ≥ 4×109/L, hemoglobin ≥ 90g/L and platelet count ≥ 100×109/L;
6. Adequate hepatic function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN) and AST or ALT ≤ 1.5 xULN;
7. Adequate renal function: creatinine clearance rate ≥ 60 ml/min or creatinine ≤ 1.5× ULN;
8. Women of childbearing potential and male participants who are sexually active must agree to use a medically effective means of birth control throughout protocol treatment;
9. Patients must be appraised of the investigational nature of the study and provide written informed consent.

Exclusion Criteria:

1. WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma;
2. Treatment with palliative intent;
3. Prior malignancy (except for adequately treated carcinoma in situ of the cervix, or basal or squamous cell carcinoma of the skin);
4. History of previous radiotherapy (except for non-melanomatous skin cancers outside intended RT treatment volume);
5. Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
6. Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period);
7. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance;
8. Prior allergic reaction to the study drug(s) involved in this protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  Defined as the time from random assignment to documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival | 2 years
  Defined as the time from random assignment to death from any cause.
Distant progression | 2 years
  Defined as the time from random assignment to the occurrence of a distant progression. Cumulative incidence of distant progression will be calculated within a competing risk framework (Fine and Gray 1999).
Locoregional progression | 2 years
  Defined as the time from random assignment to the occurrence of a locoregional progression. Cumulative incidence of locoregional progression will be calculated within a competing risk framework (Fine and Gray 1999).
Short-term response rate | 32 weeks
  Tumour response was classified according to RECIST, version 1.1
Incidence of acute and late toxicity | 2 years
  Incidence of acute toxicity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 5.0 criteria. Late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme. Acute adverse events, occurring during study treatment, and radiation-related late adverse events, occurring from 3 months after completion of radiotherapy, and chemotherapy-induced late adverse events, occurring from 3 months after completion of chemotherapy until end of follow up).

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated cancer hospital and institute of guangzhou medical university, Guangzhou, Please Select
  - Sun Yat-Sen Memorial Hospital, Guangzhou, Please Select
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Please Select
  - Dongguan people's hospital, Dongguan
  - Foshan First People's Hospital, Foshan
  - Peking university shenzhen hospital, Shenzhen
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: No